CLINICAL TRIAL: NCT06444932
Title: SUPPLEMENTARY EFFECTS OF RESISTANCE TRAINING IN ADDITION TO JOINT MOBILIZATION IN PERSONS WITH KNEE OSTEOARTHRITIS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/12
Record Dates: First submitted 2024-05-27; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Resistance Training; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Double arm parallel design RCT
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator)
  Interventions: Procedure: Joint Mobilization; Device: Transcutaneous Electric Nerve Stimulation (TENS); Device: Heating Pad
- Experimental Group (Experimental)
  Interventions: Procedure: Joint Mobilization; Procedure: Resistance Exercise Training; Device: Transcutaneous Electric Nerve Stimulation (TENS); Device: Heating Pad

INTERVENTIONS:
Procedure: Joint Mobilization — Patellofemoral and tibiofemoral joint mobilization
Procedure: Resistance Exercise Training — Lower limb resistance exercise training
  Arms: Experimental Group
Device: Transcutaneous Electric Nerve Stimulation (TENS) — Transcutaneous Electric Nerve Stimulation (TENS)
Device: Heating Pad — Heating pad for heat therapy

SUMMARY:
Joint mobilization and resistance exercise training are effective conservative treatment options for the management of osteoarthritis. However, currently no study has highlighted the supplementary effects of resistance training in addition to joint mobilization in people suffering from knee osteoarthritis. The current study is aimed at bridging the gap in literature and providing evidence regarding the additive impact of resistance training to joint mobilization in knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Knee OA grade I-III
* Individuals of either gender aged 40-70 years
* Knee OA history of no less than 3 months
* Knee pain no more than 8/10 cm on the visual analogue scale (VAS)
* Radiological evidence of grade III or less on Kellgren classification.

Exclusion Criteria:

* Those with signs of serious pathology such as malignancy, inflammatory disorder or infection.
* History of trauma or fractures in lower extremity
* Signs of lumbar radiculopathy or myelopathy
* History of knee surgery or replacement and/or receiving intra-articular steroid therapy in the preceding two months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Walking related performance fatigability | 4 weeks
  Walking related performance fatigability will be measured using 6 minute walk test. Greater fatigability indicates poorer outcome.
Stride Length | 4 weeks
  Gait analysis will be done to analyze stride length. A greater stride length signifies positive outcome and prognosis.
Gait velocity | 4 weeks
  Gait analysis will be done to analyze gaot velocity. A greater gait velocity signifies positive outcome and prognosis.
Knee Pain | 4 weeks
  Knee Pain will be measured using visual analogue scale (VAS) from 0-100mm. A higher score on VAS indicated greater pain.
Knee range of motion | 4 weeks
  Knee range of motion will be measured using a goniometer. A higher ROM signifies positive outcome.
Functional Disability | 4 weeks
  Knee functional disability will be assessed using Knee Osteoarthritis and Outcome Score (KOOS) with a score ranging from 0-100. A lower score on KOOS signifies greater functional disability.
Isometric Muscle Strength | 4 weeks
  Isometric Muscle Strength will be quantified using dynamometer. A higher score on dynamometer signifies greater muscle strength and good prognosis.
Functional capacity | 4 weeks
  5 repetition sit to stand test will be used to determine knee related functional capacity, which will be quantified in terms of time. A smaller time will denote greater functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Wania Maheen, DPT, Principal Investigator — Foundation University Islamabad; Muhammad Osama, PhD*, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation Univeristy Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No